CLINICAL TRIAL: NCT02455024
Title: A Postmarketing Observational Registry to Evaluate the Incidence of and Risk Factors for Vascular Occlusive Events Associated With ICLUSIG® (Ponatinib) in Routine Clinical Practice in the United States (OMNI).
Brief Title: An Observational Registry to Evaluate the Incidence of and Risk Factors for Vascular Occlusive Events Associated With ICLUSIG®
Acronym: OMNI
Status: Terminated | Type: Observational
Why Stopped: Business Decision; Insufficient Enrollment
Sponsor: Ariad Pharmaceuticals (Industry)
Collaborators: United BioSource, LLC (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: AP24534-14-401
Record Dates: First submitted 2015-04-17; First posted 2015-05-27 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Myeloid Leukemia, Chronic-Phase, Accelerated-Phase, Blast-Phase, Ph+ALL
Keywords: Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; ponatinib; Pharmacologic Actions; Protein Kinase Inhibitors; Risk factor; Leukemia, Myelogenous, Chronic; CML; CP-CML; Iclusig; AP24534; AP-CML; BP-CML; Ph+ALL
MeSH Terms: conditions — Leukemia, Myeloid; Blast Crisis; Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational registry to further characterize the safety profile of patients with chronic myeloid leukemia in the chronic phase (CP-CML), accelerated phase (AP-CML), blast phase (BP-CML), or Ph+ALL treated with Iclusig (ponatinib) in routine clinical practice in the US. The registry is focused on analysis of vascular occlusive events.

DETAILED DESCRIPTION:
The registry is being conducted in an effort to better understand rates, risk factors, and outcomes associated with vascular occlusive events in patients treated with Iclusig (ponatinib) in real world settings. This registry study will collect information about patient demographics, leukemia diagnosis, previous anti-cancer treatments, history of cardiovascular disease, risk factors for vascular complications, and concurrent medications (including antiplatelet and/or anticoagulant agents).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥18 years) who are diagnosed with CP-CML, AP-CML, BP-CML, or Ph+ ALL
2. Patients who are initiating Iclusig therapy for the first time, or for whom Iclusig therapy was initiated within 30 days before registry enrollment.
3. The decision to prescribe Iclusig must have been made prior to enrollment in the registry and based upon approved US indications.
4. Patients who have the ability to understand the requirements of the registry, and provide written informed consent to comply with the registry data collection procedures.

Exclusion Criteria:

1. Patients previously treated with investigational Iclusig.
2. Patients receiving any investigational agent (eg, any drug or biologic agent or medicaldevice that has not received approval in the US) or receiving Iclusig for any indication not currently approved in the US.
3. Concurrent treatment with another TKI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with CP-CML, AP-CML, BP-CML, or Ph+ALL for whom the decision to initiate treatment with commercially available Iclusig has already been made
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
The incidence of Vascular Occlusive Events (VOEs) including, but not limited to: myocardial infarction, cerebrovascular ischemic disease, peripheral artery occlusive disease and venous thromboembolism | 54 months
  All VOEs will be entered into the EDC (Electronic Data Capture system)
Number of participants with the risk factors for development of VOEs | 54 months
  Subject medical history and family medical history will be entered into the EDC
Composite outcome measure of VOEs | 54 months
  The category/type of outcome (e.g. Death, Disability/Permanent Damage, Hospitalization, Other), the time of duration, and status (continuing, resolved, fatal) will be entered into the EDC.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - John Theurer Cancer Center at Hackensack UMC (Site 128), Hackensack, New Jersey
  - Hudson Valley Hematology Oncology Associates (Site 236), Hawthorne, New York

REFERENCES:
- See also: Iclusig US Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2014/203469s009lbl.pdf
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b601a4db2bf003ab492ed??page=1&idFilter=AP24534-14-401